CLINICAL TRIAL: NCT03758573
Title: Effectiveness of Early Inspirational Muscle Training in Patients Submitted to Mechanical Ventilation: a Randomized Clinical Trial
Brief Title: Effectiveness Inspirational Muscle Training
Acronym: IMTversusMV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Rodrigo Gustavo da Silva Carvalho, Principal Investigator, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMT
Record Dates: First submitted 2018-11-21; First posted 2018-11-29 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Insufficiency
Keywords: Breathing Exercises; Respiratory Muscles; Respiration Artificial; Weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Compare the effectiveness of early inspiratory muscle training (IMT) versus non-IMT in patients undergoing mechanical ventilation to improve the outcome of mechanical ventilation weaning time.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (IMT) (Experimental): IMT by means of the Powerbreath equipment (Classic, London, UK), according to the following parameters: initial loading of 40% of MIP, 3 sets of 10 repetitions with interval of 1 minute between each sets, 7 days a week, 2 times a day , with the patients in the bed with the angulation of 45 °. The IMT load settings will be adjusted according to the values evaluated weekly. If there is need for addition of supplemental oxygen will be performed to perform the IMT.
  Interventions: Other: Inspiratory Muscle Training (IMT)
- Intensive Physiotherapy (IPT) (Active Comparator): IPT will be to individualized and supervised intervention program consisting of any of the following procedures: passive, assisted, active or resisted mobilization, sedation and orthostasis depending on the functional level of the patient, as well as bronchial hygiene therapy and pulmonary expansion therapy.
  Interventions: Other: Intensive Physiotherapy (IPT)

INTERVENTIONS:
Other: Inspiratory Muscle Training (IMT) — Inspiratory Muscle Training (IMT)
  Arms: Inspiratory Muscle Training (IMT)
Other: Intensive Physiotherapy (IPT) — Intensive Physiotherapy (IPT)
  Arms: Intensive Physiotherapy (IPT)

SUMMARY:
The long stay in mechanical ventilation can induce several complications, among them respiratory muscle weakness, this has been related to the duration of mechanical ventilation, delay and failure to wean, resulting in longer hospitalization, which reflects in greater care increase in hospital costs. Therefore, of this research will be to compare the effectiveness of early inspiratory muscle training (IMT) versus non-IMT in patients undergoing mechanical ventilation to improve the outcome of mechanical ventilation weaning time.

DETAILED DESCRIPTION:
The study will consist of a randomized controlled clinical trial conducted at the Intensive Care Unit of the University Hospital of UNIVASF. Will be included individuals of both sexes, aged 18 years or older, who are on invasive mechanical ventilation and who obtain the Free and Informed Consent Form, signed by the responsible family member. Subjects will be randomized into two groups (training and control). The inspiratory (MIP), expiratory (MEP) and peak expiratory flow pressures will be evaluated. The training group will perform respiratory muscle training, using the Powerbreath equipment, with initial loading of 40% of MIP, 7 days a week, 2 times a day. Morbidities that have repercussions on diaphragmatic contraction and end-stage disease will be used as exclusion criteria. The sample data will be analyzed through the SPSS 22.0 program. The significance level of the study will be set at 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation
* patients hemodynamically stable
* without use of vasoactive drugs

Exclusion Criteria:

* spindle trauma
* neuromuscular diseases
* end-stage disease
* pneumothorax
* rib fracture
* diaphragmatic injury
* postoperative pulmonary surgeries
* abdominal disease
* morbidities that have repercussions on diaphragmatic contraction
* mechanical ventilation with FiO2 > 60% and PEEP > 10 cm H2O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Weaning mechanical ventilation | through study completion, an average of 15 days
  time of mechanical ventilation

SECONDARY OUTCOMES:
length of stay in the ICU | through study completion, an average of 15 days
  reduction length of stay in the ICU
extubation success | through study completion, an average of 2 days
  extubation success after 48 hours
death | yes or not death, through study completion, an average of 15 days
  reduction in mortality (death)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo GS Carvalho, PhD, Principal Investigator — Physical Education College / UNIVASF
Locations (1):
- Physical Education College, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
Registration ClinicalTrials; Study Protocol; Paper results.